CLINICAL TRIAL: NCT05913986
Title: Effect of Supplementation With Alpha-lipoic Acid and Silybum Marianum (LUDLEV®) in Association With a Mediterranean Diet for the Improvement of Metabolic Dysfunction-associated Fatty Liver Disease
Brief Title: Supplementation With Alpha-lipoic Acid and Silybum Marianum(LUDLEV®) for the Improvement of Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saluz Investigación S. C. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SaluzInvestigacion
Record Dates: First submitted 2023-06-04; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Metabolic Associated Fatty Liver Disease
Keywords: fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Allocation is 1:1 to probiotic and placebo arms
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alpha-lipoic acid and y silybum marianum (Experimental): LUDLEV®300 mg/46.2 mg once day
  Interventions: Other: Placebo
- Placebo (Placebo Comparator): Placebo treatment (maltodextrin), once daily (u.i.d)
  Interventions: Dietary Supplement: LUDLEV®300 mg/46.2 mg

INTERVENTIONS:
Dietary Supplement: LUDLEV®300 mg/46.2 mg — LUDLEV®300 mg/46.2 mg once day
  Arms: Placebo
Other: Placebo — Placebo treatment (maltodextrin), once daily (u.i.d)
  Arms: Alpha-lipoic acid and y silybum marianum

SUMMARY:
This randomized, controlled, double-blind study evaluates the utility of alpha-lipoic acid and silybum marianum , versus placebo, in the treatment of metabolic associated fatty liver disease.

DETAILED DESCRIPTION:
Between 80-90% of people with associated metabolic fatty liver disease present with obesity and diabetes mellitus.

Alpha-lipoic acid is a cofactor of mitochondrial enzymes that has been considered an antioxidant since its reduced form, dihydrolipoate, reacts with reactive oxygen species and thus protects the cell membrane. Alpha-lipoic acid administration has been shown to have beneficial effects on adipokine levels and metabolic disorders such as diabetes and obesity, both of which are present in patients with MAFLD. It has been shown that the administration of 1200 mg of alpha-lipoic acid in patients with fatty liver decreases insulin resistance, serum leptin, increases the concentration of adiponectin.

Given the metabolic effects of alpha-lipoic acid, it is hypothesized that administration of this formulation may be beneficial for people with metabolic associated fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects treated at the Instituto de Investigaciones Médico Biológicas de la Universidad Veracruzana with a diagnosis of Fatty Liver Disease
* Agree to voluntarily participate in the study and sign informed consent.
* Patients with evidence of hepatic steatosis who are overweight or obese
* Patients with evidence of hepatic steatosis with diabetes mellitus and overweight or obesity.
* Patients with evidence of steatosis plus metabolic risk abnormalities will be included (waist circumference >102 in men, 88 cm in women, blood pressure >130/85 mmHg or specific treatment, triglycerides >150 mg/dL or specific treatment, HDL cholesterol < 40 mg/dL in men, <50 mg/dL in women or specific treatment, HOMA-IR >2.5, CRP >2 mg/L or prediabetes defined by fasting glucose detection 100 to 125 mg/dL, postload glucose 2 hours 140 to 199 mg/dL or HbA1c between 5.7 to 6.4%)
* Accept not to start any diet program during the study period.
* Agree not to change your current exercise plan during the study period

Exclusion Criteria:

* Patients meeting diagnostic criteria for Fatty Liver Disease with normal weight
* Patients with terminal illness, cancer, renal disease in renal replacement therapy
* Pregnant women
* Patients with inability to understand or follow the study protocol
* Sensitivity to the components of the formula.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Transitional elastography with Fibroscan | 30 minutes (performed after a 4-hour fast)

SECONDARY OUTCOMES:
controlled attenuation parameter (CAP) | 30 minutes (performed after a 4-hour fast)
  Hepatic steatosis by controlled attenuation parameter
kilopascals (kpa) | 30 minutes (performed after a 4-hour fast)
  Hepatic stiffness by Transitional elastography with Fibroscan

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Delfina Cano Contreras, Mexico, Veracruz, Mexico

DOCUMENTS (2):
  • Study Protocol (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT05913986/Prot_000.pdf
  • Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT05913986/ICF_001.pdf